CLINICAL TRIAL: NCT04159623
Title: Clinical Applicability of the Device Belk in the Rehabilitation Process
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Juan Andrés Álava, Principal Investigator, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Belk
Record Dates: First submitted 2019-11-06; First posted 2019-11-12 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Application Site Atrophy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Belk Device (Experimental): With Belk Device
  Interventions: Device: Belk Device
- Standard Rehabilitative treatment (Other): With the standard rehabilitative treatment
  Interventions: Other: Standard Rehabilitative treatment

INTERVENTIONS:
Device: Belk Device — Knee exoskeleton with electrostimulation
  Arms: Belk Device
Other: Standard Rehabilitative treatment — Use the standard rehabilitative treatment
  Arms: Standard Rehabilitative treatment

SUMMARY:
Pilot, interventional, randomized of parallel groups and multicenter clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes.
* Patients aged between 18 and 85 years.
* Patients with knee arthroplasty in the immediate postoperative period.
* Sign in informed consent.

Exclusion Criteria:

* Physical or psychological pathologies that prevent patient participation.
* Tumor arthroplasty.
* Knee replacement prosthesis.
* Impossibility of holding the device.
* Patients with a pacemaker.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
Number of sessions until recovery | An average of 12 weeks
  It is considered that the patient has completed the rehabilitation treatment when he has achieved an arc of movement between 0 and 100 degrees of flexion, a quadriceps muscle balance greater than or equal to 4/5 according to MRC (Medical Research Council)and a stable march with crutches.

SECONDARY OUTCOMES:
March in 10 meters | An average of 12 weeks
  Number of patients can be walk 10 meters
UP&Go test | An average of 12 weeks
  Do the UP&GO test
Number of falls during rehabilitation sessions | An average of 12 weeks
  Number of falls during rehabilitation sessions

CONTACTS AND LOCATIONS:
Locations (1):
- IIS Biocruces Bizkaia, Barakaldo, Bizkaia, Spain